CLINICAL TRIAL: NCT04244643
Title: Ocular Surface in Patients With Soft Contact Lenses
Acronym: E2LC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Société Française des Ophtalmologistes Adaptateurs de Lentilles de Contact (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRBN922019/CHUSTE
Record Dates: First submitted 2020-01-15; First posted 2020-01-28 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Ocular Surface
Keywords: contact lenses
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with soft contact lenses
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Data collected from patient records
  * Demographic data: date of birth, sex, city of birth
  * Contact lenses: laboratory, brand, model, wearing time before the exam, opening date of the blister, solution of contact lenses, material, renewal time
  * Refraction
  * Dry eye disease: Ocular Surface Disease Index (OSDI) score
  * LACRYDIAG data: Non-Invasive Break-Up Time (NIBUT), interferometry and tears meniscus height

SUMMARY:
Contact lenses modify the structure of the tear film by biophysical and biochemical interactions. These changes may explain more common dry eye symptoms and may sometimes cause lens failure or discontinuation.

In recent years, the investigators have various objective non-invasive methods of tear film evaluation such as the non-invasive break up time, interferometry, and tears meniscus height. These measurements are performed in clinical practice during consultation by devices such as LACRYDIAG.

The improvement of lens comfort requires a better knowledge of the ocular surface in patients with contact lenses. But currently none of these objective parameters have been accurately described.

Therefore, the investigators would like to build a database to describe the different parameters of ocular surface in patients with soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with soft contact lenses
* Patients with their contact lenses on the eyes at the time of the examination and having undergone a LACRYDIAG examination
* Only Right eye analyze

Exclusion Criteria:

* Patients with rigid contact lenses
* Patients not wearing their lenses at the time of the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft contact lenses
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
eye surface condition | baseline
  presence or not : dry eye, allergies, blepharitis, corneal abscess, corneal ulceration, corneal neovascularization, chronic inflammatory conjunctivitis and others

SECONDARY OUTCOMES:
refraction | baseline
  measured with vision tests
Ocular Surface Disease Index score | baseline
  is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.
  The overall OSDI score defined the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.
non-invasive tear break-up time | baseline
  with LACRYDIAG
interferometry | baseline
  with LACRYDIAG. Qualitative & quantitative analysis of the lipid layer.
tears meniscus height | baseline
  with LACRYDIAG

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caroline TRONE, Principal Investigator — CHU de Saint Etienne
Locations (12):
- France (12):
  - Cabinet médico-chirurgical de l'Alcazar, Beausoleil
  - Cabinet du Dr Virginie MADARIAGA, Blagnac
  - Point Vision Bordeaux, Bordeaux
  - Cabinet du Dr Françoise LE CHERPIE, Draguignan
  - Cabinet du Dr Hélène Bertrand, Lille
  - Centre ophtalmologique Saint-Paul, Paris
  - Point Vision Paris Royale, Paris
  - Centre hospitalier national d'ophtalmologie des Quinze-Vingts, Paris
  - Cabinet du Dr Cyrille TEMSTET, Paris
  - CHU de Saint Etienne, Saint-Etienne
  - Point Vision Nice - St Laurent du Var, Saint-Laurent-du-Var
  - Clinique St Jean Languedoc, Toulouse

IPD SHARING:
Plan to Share IPD: No